CLINICAL TRIAL: NCT03699007
Title: GET Living: Graded Exposure Treatment for Children and Adolescents With Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laura E Simons (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor-Investigator, Laura E Simons, Associate Professor, Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 39514; 1R21AR072921-01A1 (NIH)
Record Dates: First submitted 2018-07-28; First posted 2018-10-09 (Actual); Results first posted 2023-04-04 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Pediatric Pain; Chronic Pain, Widespread; Musculoskeletal Pain
MeSH Terms: conditions — Chronic Pain; Musculoskeletal Pain

STUDY DESIGN:
Intervention Model Description: Adolescents will be randomized to either GET Living or TPM and stratified on fear (moderate/high; FOPQ-C: moderate [35-49] high [50-96]) and disability (moderate/high; moderate [13-29] severe [30-60]), to minimize the possibility of imbalance between the two treatment arms. To allow the use of small blocks while minimizing the probability of a blinded staff member predicting the next assignment we will use blocks of size two and four and randomly choose block sizes.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Graded Exposure Therapy (GET Living) (Experimental): GET Living is jointly delivered by a pain psychologist and a physical therapist. The GET Living treatment was based on a published graded in-vivo exposure treatment manual for adults with adaptations to target a pediatric audience.
  Interventions: Behavioral: Graded Exposure Therapy (GET Living)
- Multidisciplinary Pain Management (MPM) (Active Comparator): MPM is a treatment intervention that is representative of current standards of care in a multidisciplinary pain clinic setting. It consists of Cognitive Behavioral Therapy (CBT) and Physical Therapy (PT) sessions, delivered separately by a pain psychologist and a physical therapist.
  Interventions: Behavioral: Multidisciplinary Pain Management (MPM)

INTERVENTIONS:
Behavioral: Graded Exposure Therapy (GET Living) — The protocol consists of 12 interdisciplinary sessions, 1-hour each, delivered twice a week, for an average of 6 weeks. Phase I-III are conducted with the psychologist, physical therapist, adolescent, and parent (as developmentally appropriate). Patient and parent will complete daily diaries and patients will wear the Actigraph throughout the duration of treatment.
  Arms: Graded Exposure Therapy (GET Living)
Behavioral: Multidisciplinary Pain Management (MPM) — The protocol consists of 12 multidisciplinary sessions, 1-hour each, delivered twice a week, for an average of 6 weeks. Sessions will alternate between psychological CBT sessions and Physical Therapy sessions. Patient and parent will complete daily diaries and patients will wear the Actigraph throughout the duration of treatment. The parent will also participate in 3 additional parent-only sessions with the psychologist to address parental coping skills.
  Arms: Multidisciplinary Pain Management (MPM)

SUMMARY:
The broad aim of this study is to implement and evaluate the efficacy of Graded Exposure Treatment (GET Living) to target elevated pain-related fears in children with chronic pain at the Stanford Pediatric Pain Management Clinic (PPMC). The investigators will evaluate the effectiveness and acceptability of this intervention for children with high levels of pain-related fear and functional disability. If proven efficacious, it will allow for the dissemination of this innovative treatment model to others working with children and adolescents with chronic pain.

DETAILED DESCRIPTION:
The treatment intervention to be tested in this clinical trial is Graded in-vivo Exposure Treatment (GET Living) compared to Multidisciplinary Pain Management (MPM) in adolescents with chronic musculoskeletal pain. Participants will be randomized into GET Living or MPM, and will be instructed to not seek new treatments for pain for the duration of the study. Both treatments consist of 12 1-hour patient sessions delivered twice a week across 6- weeks and 3 parent-only sessions.

ELIGIBILITY:
Inclusion Criteria:

* 8 - 18 years old; Male or Female
* Musculoskeletal pain (e.g. localized [back, limb], diffuse) not due to acute trauma (e.g. active sprain or fracture).
* Moderate to high pain-related fear ( ≥ 35 on the FOPQ-C)
* Moderate to high functional disability ( ≥ 13 on the FDI)
* English Language Proficiency

Exclusion Criteria:

* Significant cognitive impairment (e.g., brain injury)
* Significant medical or psychiatric problem that would interfere (e.g., seizures, psychosis, suicidality)

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Simons, PhD, Principal Investigator — Professor
Locations (1):
- Pediatric Pain Management Clinic - Stanford Children's Health, Menlo Park, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (text, tables, figures, appendices) that underlie the results reported in an article related to this trial will, after de-identification, be shared with researchers who provide a methodologically sound proposal.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Proposals should be directed to Dr. Laura Simons at lesimons@stanford.edu. To gain access, data requestors will need to sign a data usage agreement with Stanford University.

REFERENCES:
- [Background] Simons LE, Harrison LE, O'Brien SF, Heirich MS, Loecher N, Boothroyd DB, Vlaeyen JWS, Wicksell RK, Schofield D, Hood KK, Orendurff M, Chan S, Lyons S. Graded exposure treatment for adolescents with chronic pain (GET Living): Protocol for a randomized controlled trial enhanced with single case experimental design. Contemp Clin Trials Commun. 2019 Sep 10;16:100448. doi: 10.1016/j.conctc.2019.100448. eCollection 2019 Dec. PMID 31650069
- [Result] Shear D, Harrison LE, O'Brien S, Khazendar Z, Lyons S, Morgan JJ, Chan SK, Feinstein AB, Simons LE. Rapid Transition to Virtual Assessment and Treatment in an Interdisciplinary Randomized Clinical Trial for Youth With Chronic Pain: Adaptations and Implications for Future Trials. Clin J Pain. 2022 Jul 1;38(7):459-469. doi: 10.1097/AJP.0000000000001040. PMID 35686576
- [Derived] Simons LE, Harrison LE, Boothroyd DB, Parvathinathan G, Van Orden AR, O'Brien SF, Schofield D, Kraindler J, Shrestha R, Vlaeyen JWS, Wicksell RK. A randomized controlled trial of graded exposure treatment (GET living) for adolescents with chronic pain. Pain. 2024 Jan 1;165(1):177-191. doi: 10.1097/j.pain.0000000000003010. Epub 2023 Aug 25. PMID 37624900
- [Derived] Schemer L, Hess CW, Van Orden AR, Birnie KA, Harrison LE, Glombiewski JA, Simons LE. Enhancing Exposure Treatment for Youths With Chronic Pain: Co-design and Qualitative Approach. J Particip Med. 2023 Mar 9;15:e41292. doi: 10.2196/41292. PMID 36892929

RESULTS

PARTICIPANT FLOW:
Groups:
- Graded Exposure Therapy (GET Living): Graded Exposure Therapy (GET Living) is jointly delivered by a pain psychologist and a physical therapist: The protocol consists of 12 interdisciplinary sessions, 1-hour each, delivered twice a week, for an average of 6 weeks. Phase I-III are conducted with the psychologist, physical therapist, adolescent, and parent (as developmentally appropriate).
- Multidisciplinary Pain Management (MPM): Multidisciplinary Pain Management (MPM) protocol consists of 12 multidisciplinary sessions, 1-hour each, delivered twice a week, for an average of 6 weeks. Sessions will alternate between psychological Cognitive Behavioral Therapy (CBT) sessions and Physical Therapy sessions. The parent will also participate in 3 additional parent-only sessions with the psychologist to address parental coping skills.
Period: Treatment Phase (Baseline to 3-Month FU)
Arm/Group | Graded Exposure Therapy (GET Living) | Multidisciplinary Pain Management (MPM)
Started | 33 | 35
Completed | 26 | 33
Not Completed | 7 | 2
Not completed — Physician Decision | 7 | 2
Period: 6-month Follow Up
Arm/Group | Graded Exposure Therapy (GET Living) | Multidisciplinary Pain Management (MPM)
Started | 26 | 33
Completed | 24 | 30
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Multidisciplinary Pain Management (MPM): Multidisciplinary Pain Management (MPM) protocol consists of 12 multidisciplinary sessions, 1-hour each, delivered twice a week, for an average of 6 weeks. Sessions will alternate between psychological CBT sessions and Physical Therapy sessions. The parent will also participate in 3 additional parent-only sessions with the psychologist to address parental coping skills.
- Total: Total of all reporting groups
Arm/Group | Graded Exposure Therapy (GET Living) | Multidisciplinary Pain Management (MPM) | Total
Number analyzed (Participants) | 33 | 35 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 33 | 35 | 68
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.1 (2.92) | 14.2 (2.24) | 14.1 (2.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 24 | 55
  Male | 2 | 11 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 8 | 15
  Not Hispanic or Latino | 26 | 26 | 52
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 28 | 27 | 55
  More than one race | 0 | 4 | 4
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 33 | 35 | 68
Fear of Pain [Mean (Standard Deviation); unit: score on a scale] — Fear of Pain Questionnaire (FOPQ-C): a 24-item validated patient-report measure of pain-related fear and avoidance. The FOPQ-C contains two subscales: Fear of Pain (11 items; Min=0, Max=44) and Avoidance of Activities (13 items; Min=0, Max=52). Higher scores on each subscale indicate greater pain related fear and avoidance of activities. Here we are presenting the Fear of Pain score only.
  score on a scale | 32.36 (8.83) | 30.03 (9.59) | 31.16 (9.24)
Avoidance of Activities [Mean (Standard Deviation); unit: score on a scale] — Fear of Pain Questionnaire (FOPQ-C): a 24-item validated patient-report measure of pain-related fear and avoidance. The FOPQ-C contains two subscales: Fear of Pain (11 items; Min=0, Max=44) and Avoidance of Activities (13 items; Min=0, Max=52). Higher scores on each subscale indicate greater pain related fear and avoidance of activities. Here we are presenting the Avoidance of Activity score only.
  score on a scale | 26.67 (8.59) | 25.06 (8.71) | 25.84 (8.63)
FDI [Mean (Standard Deviation); unit: score on a scale] — Functional Disability Inventory (FDI): a 15-item validated patient-report measure of difficulties in physical, social and recreational activities (score Min=0, Max=60; Lower score means less disability/better outcome).
  score on a scale | 25.06 (10.26) | 27 (9.35) | 25.90 (9.68)

OUTCOME MEASURES:

1. Primary Outcome: Pain-related Fear and Avoidance
Description: Fear of Pain Questionnaire (FOPQ-C): a 24-item validated patient-report measure of pain-related fear and avoidance. The FOPQ-C contains two subscales: Fear of Pain (11 items; Min=0, Max=44) and Avoidance of Activities (13 items; Min=0, Max=52). Higher scores on each subscale indicate greater pain related fear and avoidance of activities.
Time Frame: Baseline to end of treatment (discharge) at 6-weeks (on average), and 3-month and 6-month follow up.
Population: Participants with data available at each time point are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Graded Exposure Therapy (GET Living) | Multidisciplinary Pain Management (MPM)
Number analyzed (Participants) | 33 | 35
score on a scale
  Fear of Pain_Baseline | 32.36 (8.83) | 30.03 (9.59)
  Fear of Pain_Discharge: number analyzed (Participants) | 27 | 33
  Fear of Pain_Discharge | 25.15 (9.14) | 25.64 (10.64)
  Fear of Pain_3 month follow-up: number analyzed (Participants) | 25 | 30
  Fear of Pain_3 month follow-up | 22.24 (11.53) | 20.03 (11.54)
  Fear of Pain_6 month follow-up: number analyzed (Participants) | 23 | 26
  Fear of Pain_6 month follow-up | 20.17 (11.25) | 21.15 (12.78)
  Avoidance of Activities_Baseline | 26.67 (8.59) | 25.06 (8.71)
  Avoidance of Activities_Discharge: number analyzed (Participants) | 27 | 33
  Avoidance of Activities_Discharge | 20.81 (8.66) | 21.61 (8.72)
  Avoidance of Activities_3 month follow-up: number analyzed (Participants) | 25 | 30
  Avoidance of Activities_3 month follow-up | 18.92 (10.75) | 18.73 (9.89)
  Avoidance of Activities_6 month follow-up: number analyzed (Participants) | 23 | 26
  Avoidance of Activities_6 month follow-up | 18.61 (10.81) | 16.77 (9.63)
Statistical Analysis 1: Comparison: Graded Exposure Therapy (GET Living) vs Multidisciplinary Pain Management (MPM); Test type: Superiority; p < 0.05, Mixed Models Analysis

2. Secondary Outcome: Functional Disability
Description: Functional Disability Inventory (FDI): a 15-item validated patient-report measure of difficulties in physical, social and recreational activities (score Min=0, Max=60; Lower score means less disability/better outcome)
Time Frame: Baseline to end of treatment (discharge) at 6-weeks (on average), and 3-month and 6-month follow up.
Population: Participants with data available at each time point are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Graded Exposure Therapy (GET Living) | Multidisciplinary Pain Management (MPM)
Number analyzed (Participants) | 33 | 33
score on a scale
  Baseline | 25.06 (10.26) | 27 (9.35)
  Discharge (approx. week 6): number analyzed (Participants) | 27 | 32
  Discharge (approx. week 6) | 20.59 (10.45) | 22 (9.58)
  3-month Follow Up: number analyzed (Participants) | 24 | 29
  3-month Follow Up | 20.08 (12.75) | 19.24 (10.08)
  6-month Follow Up: number analyzed (Participants) | 22 | 26
  6-month Follow Up | 19.82 (13.21) | 19.62 (12.28)
Statistical Analysis 1: Comparison: Graded Exposure Therapy (GET Living) vs Multidisciplinary Pain Management (MPM); Test type: Superiority; p < 0.05, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were identified from signing of ICF to end of treatment, an average duration of 6 weeks. During the 3 month and 6 month follow-up contacts, the study staff asked patient and parent if any AEs occurred since the end of treatment.
Groups:
- Typical Pain Management (TPM): Typical Pain Management (TPM) protocol consists of 12 multidisciplinary sessions, 1-hour each, delivered twice a week, for an average of 6 weeks. Sessions will alternate between psychological Cognitive Behavioral Therapy (CBT) sessions and Physical Therapy sessions. The parent will also participate in 3 additional parent-only sessions with the psychologist to address parental coping skills.
Arm/Group | Graded Exposure Therapy (GET Living) | Typical Pain Management (TPM)
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/35
Other Adverse Events (participants affected / at risk) | 0/33 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-21): https://cdn.clinicaltrials.gov/large-docs/07/NCT03699007/Prot_SAP_001.pdf
  • Informed Consent Form (2021-03-04): https://cdn.clinicaltrials.gov/large-docs/07/NCT03699007/ICF_000.pdf